CLINICAL TRIAL: NCT00126542
Title: A Phase II Trial of Bevacizumab (NSC# 704865) and OSI-774 (NSC# 718781) In Recurrent Ovarian Cancer, Fallopian Tube Carcinoma or Primary Peritoneal Carcinoma
Brief Title: Bevacizumab and Erlotinib in Treating Patients With Recurrent or Metastatic Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02660; NCI-2012-02660 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCCRC-13576A; NCI-6759; CDR0000434820; 13576A (Other: University of Chicago); 6759 (Other: CTEP); N01CM62209 (NIH); P30CA014599 (NIH); N01CM62201 (NIH); N01CM62203 (NIH)
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2012-12

CONDITIONS: Fallopian Tube Cancer; Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer; Stage IV Ovarian Epithelial Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Bevacizumab; Erlotinib Hydrochloride

ARMS (1):
- Treatment (bevacizumab, erlotinib hydrochloride) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive oral erlotinib once daily on days 1-21. Treatment repeats every 21 days for at least 3 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to 1 of the study drugs may continue treatment with the remaining study drug alone in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving bevacizumab together with erlotinib works in treating patients with recurrent or metastatic ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving bevacizumab together with erlotinib may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate in patients with recurrent or metastatic ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer treated with bevacizumab and erlotinib.

SECONDARY OBJECTIVES:

I. Determine the toxic effects of this regimen in these patients. II. Determine the median progression-free survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive oral erlotinib once daily on days 1-21. Treatment repeats every 21 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.

Patients experiencing unacceptable toxicity due to 1 of the study drugs may continue treatment with the remaining study drug alone in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer

  * Recurrent or metastatic disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable indicator lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Must have received a platinum-containing chemotherapy regimen for primary disease

  * Re-treatment with a platinum-based regimen required for patients who achieved a clinical complete response (CR) to primary therapy and then had a treatment-free interval > 12 months (i.e., platinum-sensitive) unless the patient developed a hypersensitivity to platinum

    * Patients with a treatment-free interval < 12 months do not require prior chemotherapy for recurrent disease
* No evidence of CNS disease, including primary brain tumors or brain metastasis
* Performance status - ECOG 0-2
* More than 3 months
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No history of bleeding diathesis
* SGOT and SGPT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if due to liver metastasis)
* Bilirubin normal
* INR ≤ 1.5 (3 if receiving warfarin)
* No history of esophageal varices
* Creatinine ≤ 1.5 mg/dL
* Creatinine clearance ≥ 60 mL/min
* Urine protein < 1+
* Urine protein < 1,000 mg on 24-hour urine collection
* Urine protein:creatinine ratio < 1.0
* No arterial thromboembolic event within the past 6 months, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina pectoris
  * Myocardial infarction
* No clinically significant peripheral artery disease
* No uncontrolled hypertension
* No New York Heart Association grade II-IV congestive heart failure
* No serious cardiac arrhythmia requiring medication
* No peripheral vascular disease ≥ grade 2
* Not pregnant
* No nursing during and for ≥ 3 months after study participation
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after study participation
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to study drugs (e.g., Chinese hamster ovary cell products or recombinant humanized antibodies)
* No serious or non-healing wound, ulcer, or bone fracture
* No active infection requiring parenteral antibiotics
* No other active malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No gastrointestinal tract disease resulting in an inability to take oral medication
* No significant traumatic injury within the past 28 days
* No known HIV positivity
* No prior bevacizumab
* See Disease Characteristics
* No more than 2 prior cytotoxic chemotherapy regimens for recurrent or refractory disease (i.e., failed to achieve a clinical CR after primary therapy)
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to any indicator lesion unless disease has progressed since completion of radiotherapy
* More than 4 weeks since prior major surgical procedure or open biopsy
* More than 1 week since prior core biopsy
* No prior surgery affecting absorption
* No concurrent major surgery
* Recovered from prior therapy
* No prior vascular endothelial growth factor (VEGF) or an epidermal growth factor receptor (EGFR) directed therapy
* No prior erlotinib
* At least 30 days since prior investigational drugs
* More than 1 month since prior thrombolytic agents
* Concurrent warfarin allowed provided the following criteria are met:

  * Patient is on a therapeutic stable dose of warfarin
  * INR ≤ 3
  * No active bleeding or pathological condition that would confer a high risk of bleeding (e.g., tumor invading adjacent organs or major blood vessels or varices that are likely to bleed)
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-04; Primary Completion 2007-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Response rate of patients treated with the combination of bevacizumab and OSI-774 | Up to 5 years

SECONDARY OUTCOMES:
Progression-free survival | Time from treatment commencement to disease progression or death, whichever comes first, assessed up to 5 years
  Will be analyzed using the Kaplan-Meier estimator (Kaplan 1958), and median progression-free survival times and their associated 90% confidence intervals will be determined using the method described in Brookmeyer and Crowley (Brookmeyer 1982).
Median progression-free survival | From start of treatment to time of progression, assessed up to 5 years
  Overall survival rates and median overall survival times and their associated 90% confidence intervals will be determined by the same methods.
Overall survival | Up to 5 years
  Overall survival rates and median overall survival times and their associated 90% confidence intervals will be determined by the same methods.

CONTACTS AND LOCATIONS:
Overall Officials: Gini Fleming, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States